CLINICAL TRIAL: NCT00804934
Title: Phase II Study Intravitreally Admininstered Ranibizumab in 50 Subjects With AMD Having Received at Least 3 Doses of Intermittent Anti-VEGF Therapy in the Preceding 18 Months
Brief Title: Investigates Improvement in Vision Following Switching From Avastin and Macugen Over to Lucentis
Status: Completed | Type: Observational
Sponsor: Retina Institute of Hawaii (Other)
Responsible Party: Sponsor
Other Study IDs: F4421S
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Wet AMD
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 0
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: Lucentis — 0.5mg Lucentis every four months

SUMMARY:
The purpose of this study is to determine whether people who have received intermittent anti-VEGF therapy have an improvement in vision after being switched to monthly injections of Lucentis.

DETAILED DESCRIPTION:
To determine mean change in visual acuity at 6 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age greater then and equal 50 years
* Patients with active neovascular AMD
* Received at least 3 treatments with anti-VEGF therapy (bevacizumab or pegaptanib or ranibizumab) in the last 24 months
* If the patient has bilateral disease and qualifies for the study, both eyes may be included

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from this study:
* Pregnancy or lactation
* Premenopausal women not using adequate contraception.
* Participation in another simultaneous medical investigation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-02; Primary Completion 2008-02 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Mean change in visual acuity at 6 and 12 months | one year

CONTACTS AND LOCATIONS:
Overall Officials: Debra L Shimabukuro, RN, Study Chair — Retina Institute of Hawaii
Locations (1):
- Retina Institute of Hawaii, Honolulu, Hawaii, United States